CLINICAL TRIAL: NCT03659903
Title: Long-term Benefit of Elderly Pancreatic Ductal Adenocarcinoma Patients After Pancreaticoduodenectomy
Brief Title: Pancreaticoduodenectomy in Elderly Pancreatic Ductal Adenocarcinoma Patients
Status: Completed | Type: Observational
Sponsor: The First Affiliated Hospital of Dalian Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: YJ-KY-FB-2017-06
Record Dates: First submitted 2018-09-04; First posted 2018-09-06 (Actual); Last update posted 2018-09-06 (Actual); Status verified 2018-09

CONDITIONS: Pancreas Cancer
Keywords: pancreatic ductal adenocarcinoma; pancreaticoduodenectomy
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Pancreaticoduodenectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- younger patients (age < 80): age < 80 patients， All the variables' definitions are encoded in the SEER database. To identify the PDAC cases, site codes (C25 pancreas, C25.0-C25.9) and histology codes (8140 adenocarcinoma, 8500 infiltrating duct carcinoma) based on the International Classification of Diseases for Oncology, Third Edition (ICD-O-3) were used.11 Only cases that underwent PD and microscopically confirmed were included.
  Interventions: Procedure: pancreaticoduodenectomy
- older patients (age≥ 80 ): age ≥ 80 years-old patients，All the variables' definitions are encoded in the SEER database. To identify the PDAC cases, site codes (C25 pancreas, C25.0-C25.9) and histology codes (8140 adenocarcinoma, 8500 infiltrating duct carcinoma) based on the International Classification of Diseases for Oncology, Third Edition (ICD-O-3) were used.11 Only cases that underwent PD and microscopically confirmed were included.
  Interventions: Procedure: pancreaticoduodenectomy

INTERVENTIONS:
Procedure: pancreaticoduodenectomy — pancreaticoduodenectomy

SUMMARY:
We used the SEER database to analyze the data of patients with PDAC. The database includes patients of 18 registries in the USA from 1973-2013All the malignant cases were followed-up annually to determine vital status.

The aim of Our study is to make clearly the long-term survival of younger (age <80 years) and elderly (age ≥80 years) pancreatic cancer patients underwent PD. Sec-ond, find out the risk factors of poor prognosis in elderly patients.

DETAILED DESCRIPTION:
Database We used the SEER database to analyze the data of patients with PDAC. The database includes patients of 18 registries in the USA from 1973-2013, encompassing approxi-mately 28% of the USA population. All the malignant cases were followed-up annu-ally to determine vital status.

Patient Population All the variables' definitions are encoded in the SEER database. To identify the PDAC cases, site codes (C25 pancreas, C25.0-C25.9) and histology codes (8140 adenocarcinoma, 8500 infiltrating duct carcinoma) based on the International Classification of Diseases for Oncology, Third Edition (ICD-O-3) were used.11 Only cases that underwent PD and microscopically confirmed were included.

Outcome Variables We only included those PDAC patients that underwent PD with precise data available for the following variables: age at diagnosis, year of diagnosis, gender, race, tumor site, tumor size, regional nodes positive, regional nodes examined, grade, stage, vital status, and survival months.

To clearly differentiate the difference of long-term survival between young and elderly patients, all cases were divided into two group age < 80 years and age ≥ 80 years. Since 2004, the AJCC 6th stage has been used in the SEER database. Thus, the diagnosis years of the cases included in our study ranged from 2004-2013. To analyze the median OS between different time periods, we divided the year of diagnosis into two groups: 2004-2008 year and 2009-2013. Furthermore, we also divided the tumor size into three groups: ≤ 2 cm, 2-4 cm, and > 4 cm. The lymph node ratio (LNR) is considered a robust prognostic factor after resection of pancreatic cancer and was es-timated using regional nodes positive divided by regional nodes examined.15 LNR was then categorized into three groups: 0%, 1-50%, > 50%.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pancreatic ductal adenocarcinoma，treatment by pancreaticoduodenectomy.Only cases that underwent PD and microscopically confirmed were included.

Exclusion Criteria:

* Patients with no survival data.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Pancreatic ductal adenocarcinoma patients in the SEER database form 2003 to 2013.
Sampling Method: Non-Probability Sample
Enrollment: 5910 (Actual)
Dates: Start 2004-01-01 (Actual); Primary Completion 2013-12-13 (Actual); Study Completion 2018-09-01 (Actual)

PRIMARY OUTCOMES:
median OS | to 2013 Dec. 31
  The median overall survival of all patients

IPD SHARING:
Plan to Share IPD: No